CLINICAL TRIAL: NCT07023341
Title: A Phase 3, Open Label, Single Arm Study to Evaluate Efficacy, Safety and Tolerability of Aficamten in Adult Japanese Patients With Symptomatic Obstructive Hypertrophic Cardiomyopathy
Brief Title: A Study to Learn More About How Well Aficamten Works in Japanese Participants With Symptomatic Obstructive Hypertrophic Cardiomyopathy
Acronym: CAMELLIA-HCM
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22976
Record Dates: First submitted 2025-06-10; First posted 2025-06-17 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Obstructive Hypertrophic Cardiomyopathy
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Aficamten (BAY3723113) (Experimental): Aficamten will be administered orally once daily with or without food. Participants in this arm will receive a single daily oral dose of 5 mg, 10 mg, 15 mg, or 20 mg of Aficamten with dose levels guided by echocardiography assessments, for up to 24 weeks. Participants will receive a dose of Aficamten until the drug becomes commercially available in Japan or the study ends.
  Interventions: Drug: BAY3723113

INTERVENTIONS:
Drug: BAY3723113 — Oral tablet
  Other Names: CK-3773274

SUMMARY:
Researchers are looking for a better way to treat Japanese people who have symptomatic obstructive hypertrophic cardiomyopathy (symptomatic oHCM).

Obstructive hypertrophic cardiomyopathy (oHCM) is a type of heart disease where the heart muscles become thicker than normal due to over contraction. This thickening makes it harder than normal due to over contraction. This thickening makes it harder for the heart to pump blood out to the rest of the body. In symptomatic oHCM people with the condition experience symptoms like shortness of breath, chest pain, fainting, high blood pressure and irregular heartbeats.

The study treatment aficamten, also called BAY3723113, is under development to treat symptomatic oHCM. It aims to reduce the activity of cardiac myosin, a protein that helps heart muscles to contract, and thereby preventing over contraction and muscle thickening.

Although treatment options are available for symptomatic oHCM, there is still need for other treatment options that help target the root cause of the condition. In this study, researchers want to understand about the effects and long-term safety of aficamten in Japanese people with symptomatic oHCM.

The main purpose of the study is to learn how well aficamten works in Japanese with symptomatic oCHM.

For this, the researchers will check how participant's heart blood flow changes after 6 months of treatment. They do this by measuring the pressure needed for blood to leave the heart using a test called the left ventricular outflow tract (LVOT) gradient and a special breathing technique called Valsava maneuver.

Researchers will also look for:

* the number of participants who will have at least 1 level improvement on a scale doctors use to assess the effect of heart problems on daily activities after 3 and 6 months of treatment
* the change in the impact of heart problems on participant's daily lives based on their feedback on a questionnaire called Kansas City Cardiomyopathy Questionnaire - Clinical Summary Score (KCCQ-CSS) after 3 and 6 months of treatment.

This study will have 2 treatment periods: main treatment period and long-term treatment period. During the main treatment period, participants will take aficamten tablets once daily by mouth for up to 6 months. After completing this period, the participants who can join the long-term treatment period will continue taking aficamten until the drug becomes commercially available in Japan or the study ends.

Each participant will be in the study as long as they benefit from the treatment.

Participants will visit the study site:

* once before the treatment starts
* 9 times with a gap of 2 to 4 weeks between the visits during treatment under the main treatment period, and in the long-term treatment period, participants will visit almost every 3 months until the treatment ends.
* then 2 more times with a gap of 1 month between the visits after the treatment ends.

During the study, the study doctors and their team will:

* check participant's health by performing tests such as blood and urine tests, and checking heart health using an electrocardiogram (ECG) and echocardiogram (ECHO)
* ask the participants questions about how they are feeling and what adverse events are they having

An adverse event is any medical problem that a participant has during a study. Study doctors keep track of all adverse events, irrespective if they think it is related or not to the study treatment. In addition, the participants will be asked to complete a questionnaire on quality of life at certain time points during the study.

If the participant benefits from the treatment, treatment with aficamten after the end of the study might be possible.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be 18 to 85 years of age inclusive, at the time of signing the informed consent.
* Diagnosed with HCM per the following criteria:

  1. Has LV hypertrophy and non-dilated LV chamber in the absence of other cardiac disease and
  2. Has an end-diastolic LV wall thickness as measured by the echocardiography core laboratory of:

     1. ≥15 mm in one or more myocardial segments OR
     2. ≥13 mm in one or more wall segments and a known-disease-causing gene mutation or positive family history of HCM
* Has resting LVOT-G ≥ 30 mmHg and Valsalva LVOT-G =50 mmHg during screening as determined by the echocardiography core laboratory
* LVEF ≥ 60% at screening as determined by the echocardiography core laboratory
* NYHA Functional Class II or III at screening
* Hemoglobin ≥10 g/dL at screening
* Body mass index <35 kg/m²
* Japanese
* Patients on beta-blockers, verapamil, diltiazem, or disopyramide/cibenzoline should have been on a stable regimen for >6 weeks prior to the first dose of aficamten and anticipate remaining on the same medication regimen at least during the main study treatment period. Patients treated with disopyramide or cibenzoline must also be concomitantly treated with a beta blocker and/or calcium channel blocker.

Exclusion Criteria:

* Significant valvular heart disease (per investigator judgement)

  1. Moderate-severe valvular aortic stenosis and/or regurgitation
  2. Moderate-severe mitral regurgitation not due to systolic anterior motion of the mitral valve
* Known or suspected infiltrative, genetic or storage disorder causing cardiac hypertrophy that mimics oHCM (e.g., Noonan syndrome, Fabry disease, amyloidosis)
* History of LV systolic dysfunction (LVEF <45%) or stress cardiomyopathy at any time during their clinical course
* Documented paroxysmal atrial fibrillation during the screening period
* Paroxysmal or persistent/permanent atrial fibrillation is only excluded IF:
* Rhythm restoring treatment (e.g., direct-current cardioversion, atrial fibrillation ablation procedure, or antiarrhythmic therapy) has been required ≤ 6 months prior to screening
* Rate control and anticoagulation have not been achieved for at least 6 months prior to screening
* Has been treated with SRT (surgical myectomy or percutaneous alcohol septal ablation) or cannot postpone plans for SRT until after the study period
* History of syncope or sustained ventricular tachyarrhythmia with exercise within 6 months prior to screening
* Has received prior treatment with aficamten or mavacamten

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2025-06-30 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2028-05-30 (Estimated)

PRIMARY OUTCOMES:
Change in Valsava LVOT-G | From baseline to Week 24

SECONDARY OUTCOMES:
Change in resting LVOT-G | From baseline to Weeks 12 and 24
Change in Valsava LVOT-G | From baseline to Week 12
Change in N-terminal prohormone brain natriuretic peptide (NT-proBNP) value | From baseline to Week 24
Proportion of patricipants with ≥1 class improvement in New York Heart Association (NYHA) Functional Class | From baseline to Weeks 12 and 24
Change in KCCQ-CSS score | From baseline to weeks 12 and 24
Incidence of left ventricular ejection fraction (LVEF) <40% | From baseline to last follow up, up to 4 weeks
Incidence of LVEF <50% | From baseline to last follow up, up to 4 weeks
Incidence of treatment emergent adverse events (TEAE) | From baseline to last follow up, up to 4 weeks
Incidence of treatment emergent serious adverse events (TESAE) | From baseline to last follow up, up to 4 weeks

CONTACTS AND LOCATIONS:
Locations (25):
- Japan (25):
  - Kurume University Hospital, Kurume, Fukuoka
  - Hyogo Prefectural HarimaHimeji General Medical Center, Himeji, Hyōgo
  - Kobe City Medical Center General Hospital, Kobe, Hyōgo
  - University of Tsukuba Hospital, Tsukuba, Ibaraki
  - Iwate Prefectural Central Hospital, Morioka, Iwate
  - Kitasato University Hospital, Sagamihara, Kanagawa
  - SHOWA Medical University Fujigaoka Hospital, Yokohama, Kanagawa
  - Kochi Medical School Hospital, Nankoku, Kochi
  - Mie University Hospital, Tsu, Mie-ken
  - Tohoku University Hospital, Sendai, Miyagi
  - Saiseikai Kumamoto Hospital, Kumamoto, Mumamoto
  - Kurashiki Central Hospital, Kurashiki, Okayama-ken
  - University of the Ryukyus Hospital, Ginowan, Okinawa
  - Matsushita Memorial Hospital, Moriguchi, Osaka
  - National Cerebral and Cardiovascular Center, Suita, Osaka
  - The University of Osaka Hospital, Suita, Osaka
  - Hamamatsu University Hospital, Hamamatsu, Shizuoka
  - Nippon Medical School Hospital, Bunkyo-ku, Tokyo
  - The University of Tokyo Hospital, Bunkyo, Tokyo
  - Sakakibara Heart Institute, Fuchū, Tokyo
  - Showa Medical University Koto Toyosu Hospital, Koto, Tokyo
  - Saiseikai Fukuoka General Hospital, Fukuoka
  - Gifu University Hospital, Gifu
  - Kumamoto University Hospital, Kumamoto
  - University Hospital, Kyoto Prefectural University of Medicine, Kyoto

IPD SHARING:
Plan to Share IPD: No
Currently, there is no established plan for the sharing of Individual Patient Data (IPD) from this study. The availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA 'Principles for responsible clinical trial data sharing.' This pertains to the scope, timepoint, and process of data access.
  As such, Bayer commits to considering requests from qualified researchers for patient- / study-level clinical trial data, and documents from clinical trials involving medicines and indications approved in the US and EU. However, this commitment does not reflect an active IPD sharing plan. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Researchers can use www.vivli.org to request access to IPD and documents from clinical studies to conduct research. Information on Bayer's criteria for listing studies is provided in the member section of the portal.

REFERENCES:
- See also: Click here to find further information and, after study completion, the study results according to Bayer's transparency standards. — https://clinicaltrials.bayer.com/study/22976